CLINICAL TRIAL: NCT06050798
Title: Hematological Disorder in Patients With Angiodysplasia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lydia Mamdouh Sadek Botros, Assistant lecturer, Assiut University
Other Study IDs: Angiodysplasia
Record Dates: First submitted 2023-09-16; First posted 2023-09-22 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Angiodysplasia; Hematological Disease
MeSH Terms: conditions — Angiodysplasia; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Von willebrand antigen — Von willebrand antigen change and hematological disorder in patients with angiodysplasia

SUMMARY:
The study aim will be to assess the association between GIT angiodysplasia with any hematological disorders such as any specific coagulation disorders or anemia.

DETAILED DESCRIPTION:
Angiodysplasia is a vascular GI tract abnormality tortous thin walled blood vessels seen in mucosa and submucosa highly prone to rupture resulting in GIT bleeding and hematological disorders ,Impaired coagulation profile and anemia are main changes in angiodysplasia . (An overview of angiodysplasia: management and patient prospects,Grainne Holleran et al. Expert Rev Gastroenterol Hepatol. 2018 Sep.) Gastrointestinal angiodysplasia is a major cause of recurrent bleeding. Haemostatic abnormalities have been implicated in the haemorrhage from these common vascular lesions but their precise contribution remains to be established. (Gastrointestinal angiodysplasiaG Dodda et al. J Assoc Acad Minor Phys. 1997) Angiodyplasia and aortic stenosis are both conditions that are highly prevalent in elderly people and can often co-exist. Recent studies suggest that this association is related to subtle alterations in plasma coagulation factors . The von Willebrand factor is the strongest link between aortic stenosis and bleeding associated with gastrointestinal angiodysplasia. With an aging population, the disease burden of aortic stenosis and its association with angiodysplasia of the bowel makes this an incredibly under-diagnosed yet important condition. This association when dealing with elderly patients presenting either with unexplained anemia, gastrointestinal bleeding or with aortic stenosis should be considered. A high index of suspicion and appropriate diagnostic techniques followed by appropriate and prompt treatment could be life-saving. (Heyde Syndrome Complicated by Essential Thrombocythemia: A Case Report) Chronic hematologic diseases increase the fragility of blood cell components, leading to the progressive destruction of blood cells at the site of aortic stenosis . In this process, further destruction of large multimers of von Willebrand factor may lead to coagulation disorders and gastrointestinal bleeding, such as Heyde syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adults (above 18 years) and elderly

  * Both genders
  * Admitted to GIT Unit with manifestations of GIT angiodysplasia diagnosed by upper endoscopy and Colonoscopy.
  * bleeding git symptoms

Exclusion Criteria:

* other causes ofGIT bleeding

  * bleeding git ulcers
  * hematological disorder causing bleeding tendency ex hemophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angiodysplasia
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Hematological disorder in patients with angiodysplasia | Baseline
  Von willebrand antigen change and anemia and impaired coagulation profile in angiodysplasia

CONTACTS AND LOCATIONS:
Overall Officials: AbdelHamid Mohamed AbdelHamid Aly, Study Chair — Assiut University; Nabeela Faiek Amin Mousa, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Selvam S, James P. Angiodysplasia in von Willebrand Disease: Understanding the Clinical and Basic Science. Semin Thromb Hemost. 2017 Sep;43(6):572-580. doi: 10.1055/s-0037-1599145. Epub 2017 May 5. PMID 28476066